CLINICAL TRIAL: NCT06280547
Title: Assessing the Effect of an Oral Health Education Program on Knowledge, Attitude, Practice and Dental Caries Among a Group of Children in a Governmental School in Fayoum, Egypt
Brief Title: The Effect of Oral Health Education on Knowledge, Attitude, Practice and Dental Caries Among Egyptian School Children
Acronym: KAP
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rana Hassan Ismail Ewaida, principle investigator, Cairo University
Other Study IDs: CUP 13-2; Cairo university (Other: Cairo University)
Record Dates: First submitted 2024-02-13; First posted 2024-02-28 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Dental Caries in Children; Knowledge, Attitudes, Practice
Keywords: dental caries in children; Knowledge, attitude and practice; dental caries experience; oral health education
MeSH Terms: conditions — Behavior | interventions — Health Education, Dental

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- School children aged 6-15 years old: School children aged (6 to15) years old. Children with or without previous dental experience. Children who agree to participate in the study along with a parent/guardian consent.
  Children without any mental or physical disabilities.
  Interventions: Other: Oral health education

INTERVENTIONS:
Other: Oral health education — Oral Health Education Program performed in the school.

SUMMARY:
Aim of the study Assessing the effect of an oral health education program on knowledge, attitude, practice, and dental caries among a group of school children in a governmental school in Fayoum, Egypt.

DETAILED DESCRIPTION:
Study type Others: Observational Before and after study

ELIGIBILITY:
Inclusion Criteria:

* School children aged (6 to15) years old.
* Children with or without previous dental experience.

Exclusion Criteria:

* Refusal of participation.
* Children with a mental or physical disability

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A group of Egyptian children aged between 6-15 years attending a public school in Fayoum
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2023-07-30 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
Oral health related attitude | 6 months
  Measured by close ended questionnaire, the unit of measurement is binary and the higher score is related to a positive attitude

SECONDARY OUTCOMES:
Change in oral health related Knowledge, attitude and practice | 6 months
  Measured by close ended questionnaire, the unit of measurement is binary and the higher score is related to a positive knowledge, attitude and practice accordingly

OTHER OUTCOMES:
Caries experience | 6 months
  Measured using The Caries Assessment Spectrum and Treatment (CAST) index and the unit of measurement is percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Faculty of Dentistry, Cairo, Egypt